CLINICAL TRIAL: NCT01238276
Title: Direct Antibiotic Delivery of Cefazolin Into Soft Tissue Infections Using Subcutaneous Injection and Ultrasonic Dispersion
Acronym: DAD
Status: No longer available | Type: Expanded Access
Sponsor: Sonescence, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IND 75,736
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Infection, Soft Tissue; Infection, Wound; Cellulitis; Diabetic Foot Ulcer
Keywords: soft tissue infection; wound infection; cellulitis; foot ulcer; Diabetes; antibiotics; cefazolin; cephazolin; Ancef; Kefzol; subcutaneous fluid administration; ultrasound; MRSA; Methicillin-resistant Staphylococcus aureus
MeSH Terms: conditions — Soft Tissue Infections; Wound Infection; Cellulitis; Diabetic Foot; Foot Ulcer; Diabetes Mellitus | interventions — Cefazolin

INTERVENTIONS:
Drug: Cefazolin — Cefazolin is approved for clinical use for some bacterial infections. The standard routes of administration are Intramuscular (IM) and intravenous (IV). For this study, the route of administration will be delivered using the Silberg TPS, which delivers the cefazolin by subcutaneous injection followed by external ultrasonic dispersion. The concentration delivered is one gram/100 ml saline. Cefazolin can safely be given IM at the much higher concentration of 1 gram/2.5 ml of saline. The maximum dose that may be administered is 3 grams in 300 ml, which is within the approved guidelines of a daily dose. The concentration of antibiotic will be the same; only the dose may vary depending on the size of the wound or area of induration. Each subject will receive only one treatment in this study.
  Other Names: Ancef; Kefzol
Device: Silberg Tissue Preparation System — The TPS is FDA cleared for the subcutaneous infusion and ultrasonic dispersion of tumescent fluid excluding the parenteral delivery of drugs. Under this study, the TPS is a device to deliver cefazolin by subcutaneous injection followed by external ultrasonic dispersion. The TPS consists of a medical grade peristaltic pump that is used to infuse antibiotic solution using a sterile blunt-tipped infusion cannula into a superficial subcutaneous plane. After the cannula has been removed, high frequency external ultrasound is delivered transcutaneously over the area of infusion in order to disperse the antibiotic solution. The power density is within the range allowed for physical therapy.
  Other Names: Silberg TPS (K023083); Tissue Preparation System; TPS; Mettler ME800

SUMMARY:
This study focuses on a new drug delivery system (Direct Antibiotic Delivery) to treat soft tissue infections. In this study, cefazolin is delivered directly to the target tissues using subcutaneous injection of antibiotic solution and then dispersed using high-frequency external ultrasound. Using this system, a much higher concentration of antibiotic can be achieved than through traditional treatment methods.

Unlike traditional delivery methods, Direct Antibiotic Delivery does not rely on blood supply and is beneficial for subjects with Diabetes or subjects who have received radiation therapy and blood supply is limited.

DETAILED DESCRIPTION:
In this study, the DOSAGE of cefazolin that is delivered is a fraction of that which is already FDA approved for intramuscular (IM) administration. However, the CONCENTRATION in the target area is much higher than what can be achieved through intravenous (IV) administration, while still being far less than what is approved for IM administration.

Previous to this study, cefazolin was considered to be ineffective in treating Methicillin-resistant Staphylococcus aureus (MRSA) as it had only been tested at the concentrations that were attainable by traditional methods. Through our study and laboratory tests conducted at the Harford Hospital, Connecticut, we have confirmed that cefazolin can be effective against even the most resistant strains of MRSA if a high enough concentration is obtained.

Under this study, treatment is only available to subjects that have already undergone standard therapy, but were not able to resolve the infection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pathologically confirmed presence of serious or immediately life-threatening soft tissue infection, cellulitis or open wound caused by bacteria for which cefazolin at this concentration is likely to have activity to inhibit the bacteria, for example, Staphylococcus species or Streptococcus species, Escherichia coli, Proteus mirabilis.
* Wounds must demonstrate the presence of skin and skin structure infection, which may be demonstrated by one or more of the following: Culture results as aforementioned, swelling of the tissues, discoloration, open wounds, and/or drainage, which may or may not be associated with pain and/or tenderness.
* Confirmed presence of soft tissue cellulitis caused by bacteria for which cefazolin is likely to have activity to inhibit the bacteria will be evidenced by microbiologic cultures taken no greater than ten (10) days prior to treatment.
* Subject must have previously been treated by a qualified licensed physician using traditional surgical and/or medical treatments, which may include courses of IV antibiotics, but where Subject was unable to resolve their infection through traditional surgical and/or medical treatments for soft tissue cellulitis caused by bacteria for which cefazolin is likely to have activity to inhibit the bacteria at a maximum concentration of 1 gram per 100 ml saline, as demonstrated by the presence of induration, redness, open wounds, and/or soft tissue swelling.
* Subject must be referred by his or her treating physician to the Wound Care Center of the investigational hospital.
* The Wound Care Center of the investigational hospital has confirmed that standard therapies have failed to cure the subject's infection and the infection is still present.
* Subjects are not on concomitant antibacterial drugs since these drugs have failed to treat the subject's infection.
* Subject may be male or female and must be at least 18 years of age.
* Subject must sign informed consent as approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* Subjects who have not received treatment by traditional surgical and/or medical therapies.
* Subjects who are allergic to cefazolin.
* Subjects who have a serious allergy to penicillin.
* Subjects with infections that involve body cavities.
* Subjects designated to be vulnerable, i.e., pregnant women, subjects under the age of 18, and subjects who need to have consent provided by a Legally Authorized Representative (LAR).
* Subjects who are unable or unwilling to comply with the protocol.
* Subjects who have a history of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association (NYHA) functional classification of 3.
* Subjects who have any other life-threatening illness or organ system dysfunction, which, in the opinion of the investigator, would either compromise subject safety or interfere with the evaluation of the safety of the test drug.
* Subjects who cannot understand English.
* Subjects who have received a treatment under this study are not eligible for re-admittance for thirty (30) days from the date of their last treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Barry N Silberg, MD, Principal Investigator — Sonoma West Medical Center, Santa Rosa Memorial Hospital, Sutter Health; James K Gude, MD, Study Director — Sonoma West Medical Center
Locations (1):
- Sonoma West Medical Center, Sebastopol, California, United States

REFERENCES:
- [Background] Weninger KR, Camara CG, Putterman SJ. Observation of bubble dynamics within luminescent cavitation clouds: Sonoluminescence at the nano-scale. Phys Rev E Stat Nonlin Soft Matter Phys. 2001 Jan;63(1 Pt 2):016310. doi: 10.1103/PhysRevE.63.016310. Epub 2000 Dec 27. PMID 11304356
- [Background] Lavery LA, Armstrong DG, Murdoch DP, Peters EJ, Lipsky BA. Validation of the Infectious Diseases Society of America's diabetic foot infection classification system. Clin Infect Dis. 2007 Feb 15;44(4):562-5. doi: 10.1086/511036. Epub 2007 Jan 17. PMID 17243061
- [Background] Frisoli Junior A, de Paula AP, Feldman D, Nasri F. Subcutaneous hydration by hypodermoclysis. A practical and low cost treatment for elderly patients. Drugs Aging. 2000 Apr;16(4):313-9. doi: 10.2165/00002512-200016040-00007. PMID 10874526
- [Background] Champoux N, Du Souich P, Ravaoarinoro M, Phaneuf D, Latour J, Cusson JR. Single-dose pharmacokinetics of ampicillin and tobramycin administered by hypodermoclysis in young and older healthy volunteers. Br J Clin Pharmacol. 1996 Sep;42(3):325-31. doi: 10.1046/j.1365-2125.1996.03967.x. PMID 8877023